CLINICAL TRIAL: NCT06608992
Title: Evaluation of the Safety and Hemostatic Effectiveness of SURGICEL® Powder in TKA：a Randomized Controlled Trial
Brief Title: Evaluation of the Effect of SURGICEL® Powder in TKA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP-TKA-RCT
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-09

CONDITIONS: Knee Osteoarthritis
Keywords: total knee arthroplasty; knee osteoarthritis; SURGICEL® Powder; the safety and hemostatic effectiveness
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: According to the inclusion/exclusion criteria for study participants, patients undergoing unilateral primary total knee arthroplasty will be screened. After obtaining informed consent from the patients, computer-based randomization will be conducted. The patients included in the study will be randomly assigned to either the test group (using SURGICEL® Powder ) or the control group (not using SURGICEL® Powder ).
Who Masked: Participant, Investigator
Masking Description: During the trial, patients will not be aware of which hemostatic method corresponds to their assigned group. Except for the operating surgeon, the perioperative assessment of various parameters for the patients will be conducted by a medical team that is also unaware of the intraoperative hemostatic method used for the patient. Thus, the study achieves both patient blinding and assessor blinding, except for the surgeon. Unblinding will occur after the finalization of the statistical analysis plan, data audit report, and database lock, at which point the group assignment corresponding to the treatment group will be revealed. In emergency situations, if the researcher believes that revealing the intraoperative method used would benefit the handling of adverse events, emergency unblinding may occur.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- using SURGICEL® Powder (Experimental): The SURGICEL® Powder will be sprayed in areas such as the posterior joint capsule, medial gap, lateral gap, suprapatellar pouch, and infrapatellar fat pad. After the SURGICEL® Powder fully react and change color, any unreacted SURGICEL® Powder will be appropriately washed using an irrigation gun.
  Interventions: Drug: SURGICEL® Powder
- not using SURGICEL® Powder (No Intervention): The SURGICEL® Powder will not be used during the surgery.

INTERVENTIONS:
Drug: SURGICEL® Powder — SURGICEL® Powder are hemostatic product made of compacted, regenerated oxidized cellulose fine fiber aggregates, produced using a patented process. These particles are pre-loaded into an applicator device for application to the target bleeding site. SURGICEL® Powder are white with a slight yellow tint and have a faint caramel-like scent.When SURGICEL® Powder are fully saturated with blood, they expand into a brown or black gel-like substance that helps form a blood clot. This substance acts as a hemostatic adjunct to control localized bleeding.
  Arms: using SURGICEL® Powder

SUMMARY:
The study subjects are patients in our hospital's orthopedics department undergoing unilateral primary total knee arthroplasty (TKA) due to primary osteoarthritis. Through a prospective, parallel randomized controlled study, 112 participants will be divided into two groups: the SURGICEL® Powder group and the non-use group. The study will compare the total perioperative blood loss , intraoperative blood loss, transfusion rate and volume, postoperative hemoglobin decline, hematocrit decline, limb swelling rate , postoperative limb pain , and range of motion. Statistical analysis will be performed on the data to observe the hemostatic effects of SURGICEL® Powder, providing recommendations for the clinical use of SURGICEL® Powder.

DETAILED DESCRIPTION:
The study subjects are patients in our hospital's orthopedics department undergoing unilateral primary total knee arthroplasty (TKA) due to primary osteoarthritis. Through a prospective, parallel randomized controlled study, 112 participants will be divided into two groups: the SURGICEL® Powder group and the non-use group. The study will compare the total perioperative blood loss (on postoperative days 3 and 5), intraoperative blood loss, transfusion rate and volume, postoperative hemoglobin decline, hematocrit decline, limb swelling rate (postoperative days 1-5), postoperative limb pain (measured by the Visual Analogue Scale, VAS, on days 1-5), and range of motion (ROM on days 1-5). Statistical analysis will be performed on the data to observe the hemostatic effects of SURGICEL® Powder, providing recommendations for the clinical use of SURGICEL® Powder.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with primary knee osteoarthritis based on symptoms, physical examination, and imaging, with X-ray showing Kellgren-Lawrence (K-L) stage III or higher.
2. Severe knee pain with functional limitations, unresponsive to conservative treatment, and scheduled for unilateral primary total knee arthroplasty (TKA).
3. No severe knee deformity (flexion deformity >30°, varus >20°, or valgus >10°).
4. Patients undergoing manual surgery with traditional instruments.

Exclusion Criteria:

1. History of long-term anticoagulant use for more than 3 months due to cardiovascular or cerebrovascular disease and failure to stop medication (Aspirin/Clopidogrel <7 days, Warfarin <5 days, or Reserpine <7 days), or the presence of the following conditions: renal insufficiency (blood urea nitrogen ≥25.3 mmol/L or serum creatinine ≥442 μmol/L), liver insufficiency (ALT or AST ≥80 U/L), severe heart disease (or coronary stent placement within the last 12 months), severe respiratory disease (lung function FEV1.0 <0.5L or FEV1.0/FVC <60%), history of venous thromboembolism (VTE) or high risk of thrombosis (hereditary/acquired thrombotic disorders), coagulation disorders (APTT ≥46 seconds or INR ≥1.7), stroke, or history of malignant tumors; anemia (according to WHO anemia diagnosis criteria, Hb <130 g/L for males and <120 g/L for females).
2. Patients undergoing TKA surgery with the assistance of robotic or navigation digital technology.
3. Presence of other contraindications to total knee arthroplasty, such as metal allergies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-09-28 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
total perioperative blood loss | 1 day after surgery
  Total Blood Loss = Preoperative Blood Volume (PBV) × (Preoperative Hematocrit - Postoperative Hematocrit) / Average Hematocrit + Transfusion Volume
  Where:
  Average Hematocrit = (Preoperative Hematocrit + Postoperative Hematocrit) / 2
  PBV is calculated using Nadler's method:
  PBV = K1 × Height (m)³ + K2 × Weight (kg) + K3 For males: K1 = 0.3669, K2 = 0.03219, K3 = 0.6041 For females: K1 = 0.3561, K2 = 0.03308, K3 = 0.1833；The lower it is, the better the hemostatic effect.
total perioperative blood loss | 2 days after surgery
  Total Blood Loss = Preoperative Blood Volume (PBV) × (Preoperative Hematocrit - Postoperative Hematocrit) / Average Hematocrit + Transfusion Volume
  Where:
  Average Hematocrit = (Preoperative Hematocrit + Postoperative Hematocrit) / 2
  PBV is calculated using Nadler's method:
  PBV = K1 × Height (m)³ + K2 × Weight (kg) + K3 For males: K1 = 0.3669, K2 = 0.03219, K3 = 0.6041 For females: K1 = 0.3561, K2 = 0.03308, K3 = 0.1833；The lower it is, the better the hemostatic effect.
total perioperative blood loss | 3 days after surgery
  Total Blood Loss = Preoperative Blood Volume (PBV) × (Preoperative Hematocrit - Postoperative Hematocrit) / Average Hematocrit + Transfusion Volume
  Where:
  Average Hematocrit = (Preoperative Hematocrit + Postoperative Hematocrit) / 2
  PBV is calculated using Nadler's method:
  PBV = K1 × Height (m)³ + K2 × Weight (kg) + K3 For males: K1 = 0.3669, K2 = 0.03219, K3 = 0.6041 For females: K1 = 0.3561, K2 = 0.03308, K3 = 0.1833；The lower it is, the better the hemostatic effect.
total perioperative blood loss | 4 days after surgery
  Total Blood Loss = Preoperative Blood Volume (PBV) × (Preoperative Hematocrit - Postoperative Hematocrit) / Average Hematocrit + Transfusion Volume
  Where:
  Average Hematocrit = (Preoperative Hematocrit + Postoperative Hematocrit) / 2
  PBV is calculated using Nadler's method:
  PBV = K1 × Height (m)³ + K2 × Weight (kg) + K3 For males: K1 = 0.3669, K2 = 0.03219, K3 = 0.6041 For females: K1 = 0.3561, K2 = 0.03308, K3 = 0.1833；The lower it is, the better the hemostatic effect.
total perioperative blood loss | 5 days after surgery
  Total Blood Loss = Preoperative Blood Volume (PBV) × (Preoperative Hematocrit - Postoperative Hematocrit) / Average Hematocrit + Transfusion Volume
  Where:
  Average Hematocrit = (Preoperative Hematocrit + Postoperative Hematocrit) / 2
  PBV is calculated using Nadler's method:
  PBV = K1 × Height (m)³ + K2 × Weight (kg) + K3 For males: K1 = 0.3669, K2 = 0.03219, K3 = 0.6041 For females: K1 = 0.3561, K2 = 0.03308, K3 = 0.1833；The lower it is, the better the hemostatic effect.

SECONDARY OUTCOMES:
pain visual analogue scale score | 1 day after surgery
  pain visual analogue scale score; range from 0 to 10; The lower it is, the better the analgesic effect
pain visual analogue scale score | 2 days after surgery
  pain visual analogue scale score; range from 0 to 10; The lower it is, the better the analgesic effect
pain visual analogue scale score | 3 days after surgery
  pain visual analogue scale score; range from 0 to 10; The lower it is, the better the analgesic effect
pain visual analogue scale score | 4 days after surgery
  pain visual analogue scale score; range from 0 to 10; The lower it is, the better the analgesic effect
pain visual analogue scale score | 5 days after surgery
  pain visual analogue scale score; range from 0 to 10; The lower it is, the better the analgesic effect
pain visual analogue scale score | 2 weeks after surgery
  pain visual analogue scale score; range from 0 to 10; The lower it is, the better the analgesic effect
Limb Swelling Rate | Postoperative day 1
  (Postoperative circumference 10 cm above the patella - Preoperative circumference 10 cm above the patella) / Preoperative circumference 10 cm above the patella.
Limb Swelling Rate | Postoperative day 2
  (Postoperative circumference 10 cm above the patella - Preoperative circumference 10 cm above the patella) / Preoperative circumference 10 cm above the patella.
Limb Swelling Rate | Postoperative day 3
  (Postoperative circumference 10 cm above the patella - Preoperative circumference 10 cm above the patella) / Preoperative circumference 10 cm above the patella.
Limb Swelling Rate | Postoperative day 4
  (Postoperative circumference 10 cm above the patella - Preoperative circumference 10 cm above the patella) / Preoperative circumference 10 cm above the patella.
Limb Swelling Rate | Postoperative day 5
  (Postoperative circumference 10 cm above the patella - Preoperative circumference 10 cm above the patella) / Preoperative circumference 10 cm above the patella.
Coagulation Testing | Postoperative day 1
  Assay index including D-dimers and Activated partial thromboplastin time.
Coagulation Testing | Postoperative day 2
  Assay index including D-dimers and Activated partial thromboplastin time.
Coagulation Testing | Postoperative day 3
  Assay index including D-dimers and Activated partial thromboplastin time.
Coagulation Testing | Postoperative day 4
  Assay index including D-dimers and Activated partial thromboplastin time.
Coagulation Testing | Postoperative day 5
  Assay index including D-dimers and Activated partial thromboplastin time.
Knee range of motion | Postoperative day 1
  The rehabilitation doctor takes the measurements of changes in knee joint motion during the first three days after surgery
Knee range of motion | Postoperative day 2
  The rehabilitation doctor takes the measurements of changes in knee joint motion during the first three days after surgery
Knee range of motion | Postoperative day 3
  The rehabilitation doctor takes the measurements of changes in knee joint motion during the first three days after surgery
Knee range of motion | Postoperative day 4
  The rehabilitation doctor takes the measurements of changes in knee joint motion during the first three days after surgery
Knee range of motion | Postoperative day 5
  The rehabilitation doctor takes the measurements of changes in knee joint motion during the first three days after surgery
Knee range of motion | Postoperative day 14
  The rehabilitation doctor takes the measurements of changes in knee joint motion during the first three days after surgery
Blood routine | Postoperative day 1
  Assay index including white blood cell count and neutrophil count.
Blood routine | Postoperative day 2
  Assay index including white blood cell count and neutrophil count.
Blood routine | Postoperative day 3
  Assay index including white blood cell count and neutrophil count.
Blood routine | Postoperative day 4
  Assay index including white blood cell count and neutrophil count.
Blood routine | Postoperative day 5
  Assay index including white blood cell count and neutrophil count.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Tian, doctor, Study Chair — Director
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No